CLINICAL TRIAL: NCT04309825
Title: Efficacy of Transgastrostomal Esophagogastroduodenoscopies in Children
Brief Title: Transgastrostomal Endoscopies
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no IRB approval
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000027348
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Esophagogastroduodenoscopies

STUDY DESIGN:
Intervention Model Description: To examine the efficacy of transgastrostomal endoscopies among a single group of patients with a gastrostomy feeding tube
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- G-tube endoscopies patients (Experimental): patients who will undergo an endoscopy through g-tube port
  Interventions: Procedure: transgastrostomal endoscopy

INTERVENTIONS:
Procedure: transgastrostomal endoscopy — Placement the endoscope through the g-tube port and not through the mouth of a patient undergoing an upper gi endoscopy

SUMMARY:
Upper GI endoscopies are commonly done by inserting the endoscope through the patient's mouth. When a patient has a gastrostomy feeding tube, the endoscope can be inserted through the stomach port opening. The aim is to prove this modification would lead to various health benefits, including need for lighter anesthesia, rapid recovery time and fewer anesthesia related adverse reactions.

DETAILED DESCRIPTION:
Pediatric esophagogastroduodenoscopies (EGD) are commonly used for diagnosis and treatment of various GI conditions. Appropriate sedation or anesthesia and analgesia is critical for enhancing the effectiveness and feasibility of EGD. General anesthesia or deep sedation are commonly used for this procedure. Midazolam is the most common intravenous sedative in use, often in combination with ketamine, propofol, meperidine or fentanyl.

Despite technical advances in patient monitoring and the safety of anesthesia and sedation drugs, procedural anesthesia or sedation adverse events may occur. Desaturation during the procedure is the most common adverse event, followed by vomiting, excessive secretion and unexpected apnea. Children with aero-digestive pathologies and feeding disorders often carry significant underlying co-morbidities, increasing their anesthesia risk. Previous studies have shown that caution must be exercised in children with potential airway problems or uncorrected cardiopulmonary anomalies such as laryngomalacia, chromosomal abnormalities, tetralogy of fallot and bronchopulmonary dysplasia. In addition, this population is often at increased risk for concurrent respiratory conditions, which may increase the risk for laryngospasm during the procedure.

As the endoscope is inserted transorally, it may also be an important trigger for laryngospasm. Alternatives to oral insertion of the endoscope have been described and shown to be more beneficial than the oral route in some patients. For example, previous studies have shown that transnasal endoscopies are known to be less of a burden to patients, and have benefits including fewer effects on respiratory and cardiovascular status and reduced recovery time after procedure.

Alternatively, insertion of the endoscope through the gastrocutaneous tract is possible among patients with a percutaneous gastrostomy feeding tube. This technique has been well described in the adult population for observation, diagnosis and treatment of various digestive diseases. As children with aero-digestive and feeding disorders often have a percutaneous gastrostomy feeding tube, and are at increased risk for anesthesia adverse events, transgastrostomal endoscopies me be beneficial in this patient population. To date, this method has not been reported and examined in children undergoing EGDs.

The aims of this study:

1. Examine the feasibility of transgastrostomal EGDs in children Assess the ability to explore the upper GI tract from proximal esophagus to the second part of the duodenum and obtain adequate tissue biopsies.
2. Assess the need for anesthesia and sedation In the adult population transgastrostomal endoscopies are done with no anesthesia or sedation. Previous studies on adult population have shown that even with lack of sedation, this procedure was not associated with any decrease of oxygen saturation nor a significant difference in fluctuations of blood pressures and heart rate in comparison to oral EGDs. As for children, a "lighter" anesthesia with inhalation with a face mask or sedation with intranasal application of dexmedetomidine hydrochloride may provide adequate anesthesia or sedation for this procedure. However, the decision regarding the type of anesthesia used during endoscopy remains per anesthesiologist discretion and is not part of this study.
3. Examine the benefits of this procedure in comparison to oral EGD Specifically, will examine the rate of procedural sedation or anesthesia adverse events and patients' recovery time.

4. Research Plan:

Study will take place at the children's operating room of Yale New Haven Hospital.

Enrollment to the study will take place on the day of the endoscopy during the pre-procedural assessment. Eligible patients will be offered to have a transgastrostomal endoscopy instead of a transoral one.

Similar to a transoral EGD, on the patient's arrival to the operating room (OR) the anesthesia team will obtain vital signs (blood pressure, heart rate, respiratory rate and oxygen saturation). Those would be monitored continuously during the procedure.

Once the preprocedural assessment is completed, the anesthesiologist will determine the type of anesthesia: intravenous drugs, gas inhalation or intranasal dexmedetomidine hydrochloride at a standard dosage of 2 mcg/kg. As "lighter" anesthesia may be used in this study (compared to transoral EGDs), the depth of anesthesia will be continuously monitored. The patients will be connected to a bispectral index (BIS) monitor, which identifies changes in electrophysiologic brain activity during general anesthesia. The BIS monitor, derived from electroencephalogram (EEG) data, has been shown to be a useful cerebral monitor of anesthesia depth.

Once the patient is laid in the supine position, the gastrostomy tube is removed. After applying a lubricant around the endoscope, it is inserted through the fistural tract and advanced into the gastric lumen. At this point a standard endoscopy will be conducted (with no significant changes compared to a transoral EGD). The endoscope is directed to the oral side and advanced to the esophagogastric junction. The endoscope is retrogradely inserted through the esophagus, and proximal and distal esophageal biopsies are obtained. The endoscope is then withdrawn to the stomach and directed to the anal side. The endoscope is inserted up to the second part of the duodenum from the stoma. Duodenal biopsies are obtained from the 2nd duodenal part and the duodenal bulb. The endoscope is pulled back to the stomach and turned back to look around the stoma. Gastric biopsies are obtained from the body of the stomach and the pre-pyloric region. After observation of the upper gastrointestinal tract, air is suctioned and the endoscope is withdrawn from the stoma. The gastrostomy tube is placed.

Procedure length is estimated at 15 minutes.

The main differences between a standard transoral endoscopy and a trandgastrotsotmal one are:

1. Insertion of the endoscope through the G-tube port and not the mouth.
2. The need to remove the existing G-tube and replace it once the endoscopy is done
3. Potential use of "lighter" sedation. In this study the depth of anesthesia will be monitored with a BIS monitor. This monitor is not used during a standard EGD.

The procedure's efficacy, length and adverse reaction will be compared to the standard transoral endoscopy.

ELIGIBILITY:
Inclusion Criteria:

- children with a percutaneous gastrostomy feeding tube, who are about to have a diagnostic esophagogastroduodenoscopy.

Exclusion Criteria:

* age>18 years,
* G-tube size <12Fr.
* Patients with immature gastrocutaneous fistula (< 4 weeks after gastrostomy)

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Obtain adequate biopsies | 15 minutes
  Conduct a full endoscopy via g-tube port. Advance the scope to all standard locations including proximal esophagus, distal esophagus, stomach, duodenal bulb and the second part of the duodenum. Obtain at least 2 specimens from each location.

SECONDARY OUTCOMES:
anesthesia related adverse reactions | 15 minutes
  Assess the rate of anesthesia related adverse reactions. Specifically, record the number of oxygen desaturations during the endoscopy (vital signs are continuously recorded during the exam). After the procedure the anesthesia team will summarize any anesthesia adverse reactions that have occurred during the exam.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedt M, Welsch S. An update on pediatric endoscopy. Eur J Med Res. 2013 Jul 25;18(1):24. doi: 10.1186/2047-783X-18-24. PMID 23885793
- [Background] van Beek EJ, Leroy PL. Safe and effective procedural sedation for gastrointestinal endoscopy in children. J Pediatr Gastroenterol Nutr. 2012 Feb;54(2):171-85. doi: 10.1097/MPG.0b013e31823a2985. PMID 21975965
- [Background] Campo R, Montserrat A, Brullet E. Transnasal gastroscopy compared to conventional gastroscopy: a randomized study of feasibility, safety, and tolerance. Endoscopy. 1998 Jun;30(5):448-52. doi: 10.1055/s-2007-1001306. PMID 9693891
- [Background] Dumortier J, Ponchon T, Scoazec JY, Moulinier B, Zarka F, Paliard P, Lambert R. Prospective evaluation of transnasal esophagogastroduodenoscopy: feasibility and study on performance and tolerance. Gastrointest Endosc. 1999 Mar;49(3 Pt 1):285-91. doi: 10.1016/s0016-5107(99)70002-7. PMID 10049409
- [Background] Mori A, Ohashi N, Maruyama T, Tatebe H, Sakai K, Shibuya T, Inoue H, Takegoshi S, Okuno M. Transnasal endoscopic retrograde chalangiopancreatography using an ultrathin endoscope: a prospective comparison with a routine oral procedure. World J Gastroenterol. 2008 Mar 14;14(10):1514-20. doi: 10.3748/wjg.14.1514. PMID 18330940
- [Background] Adler DG, Gostout CJ, Baron TH. Percutaneous transgastric placement of jejunal feeding tubes with an ultrathin endoscope. Gastrointest Endosc. 2002 Jan;55(1):106-10. doi: 10.1067/mge.2002.119257. PMID 11756929